CLINICAL TRIAL: NCT03398759
Title: Butorphanol Mitigate Emergence Agitation in Patients Undergoing Functional Endoscopic Sinus Surgery：a Randomized Control Double Blinded Clinical Trail
Brief Title: Butorphanol Mitigate Emergence Agitation in Patients Undergoing Functional Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Xiaorong Huai, resident physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FNPA2017
Record Dates: First submitted 2018-01-03; First posted 2018-01-12 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Agitation
Keywords: Butorphanol; Functional endoscopic sinus surgery; Emergence agitation
MeSH Terms: conditions — Psychomotor Agitation; Emergence Delirium | interventions — Butorphanol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butorphanol (Experimental): Butorphanol 20ug/kg , anesthesia induction，Intravenous injection
  Interventions: Drug: Butorphanol
- Placebo (Placebo Comparator): Normal saline 5ml ， anesthesia induction，Intravenous injection
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Butorphanol — IV injection during induction
  Arms: Butorphanol
Drug: Placebos — IV injection during induction
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Emergence agitation is one of the common postoperative complications after functional endoscopic sinus surgery（FESS). The objective of present study is to explore the effectiveness of butorphanol in the alleviation of emergence agitation in patients undergoing Functional Endoscopic Sinus Surgery.

DETAILED DESCRIPTION:
Butorphanol is a mixed agonist-antagonist opioid with strong κappa-receptor agonist and weak mu-receptor antagonist activity. It is commonly used for the management of cancer, postoperative, gynecologic, and obstetric pain. Additionally, Butorphanol has less respiratory depression and sedation effects, which make it may become a good medicine to alleviate the agitation. However, there is no clinical evidence to confirmation of such effectiveness of butorphanol. The objective of present study is to explore the effectiveness of butorphanol in the alleviation of emergence agitation in patients undergoing Functional Endoscopic Sinus Surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years,<=65years;
2. height 150-180 cm;
3. weight 55-80 kg;
4. Signed the inform consent
5. American Society of Anesthesiologists classification I to II
6. Select to functional endoscopic sinus surgery

Exclusion Criteria:

1. Existing cerebral disease, or have a history of neurological and psychiatric diseases including Alzheimer Disease, stroke, epilepsy and psychosis;
2. Several audition or vision disorder;
3. Unwillingness to comply with the protocol or procedures.
4. Can not communicated with Chinese Mandarin
5. Existing bradycardiac arrhythmia（Heart rate <60 bpm for any reasons）
6. Existing gastrointestinal ulcer
7. Existing urinary incontinence
8. Existing asthma or chronic obstructive pulmonary disease
9. Allegory to Butorphanol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Emergence agitation incidence | 1 hour in the post anesthesia care unite(PACU)
  Emergence agitation incidence

SECONDARY OUTCOMES:
MAP | 1 hour in the post anesthesia care unite(PACU)
  The mean arterial pressure
HR | 1 hour in the post anesthesia care unite(PACU)
  Heart rate
quality of recovery -40 questionnaire | 24h after operation
  Measurement of quality of recovery with QoR-40

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, MD, Study Chair — Anesthesiology Department Renji Hospital, Shanghai
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang X, Qi S, Lin Z, Zhang Y, Dai W, Tian W, Tian J, Zheng L, Su D, Huai X. Pre-operative administration of butorphanol mitigates emergence agitation in patients undergoing functional endoscopic sinus surgery: A randomized controlled clinical trial. Front Psychiatry. 2023 Jan 17;13:1090149. doi: 10.3389/fpsyt.2022.1090149. eCollection 2022. PMID 36733413